CLINICAL TRIAL: NCT01068613
Title: A Randomized, Double-blind, Double-dummy, Three Period Incomplete Cross-over Study to Evaluate the Safety and Efficacy of Multiple Daily Doses of QAX028 as Compared to Tiotropium Bromide (Positive Control) and Placebo in COPD Patients
Brief Title: Safety and Efficacy of Multiple Doses of QAX028 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAX028A2201
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Long acting muscarinic antagonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- QAX028 high dose (Experimental)
  Interventions: Drug: QAX028
- QAX028 low dose (Experimental)
  Interventions: Drug: QAX028
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAX028 — QAX028 60 mcg via inhalation device
  Arms: QAX028 high dose
Drug: QAX028 — QAX028 20 mcg via inhalation device
  Arms: QAX028 low dose
Drug: Tiotropium — Tiotropium via inhalation device
  Arms: Tiotropium
Drug: Placebo — Placebo to QAX028 via inhalation device
  Arms: Placebo

SUMMARY:
This study will assess the bronchodilator effects of multiple doses of QAX028 at two different dose levels when compared to tiotropium and placebo in a COPD population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to GOLD guidelines
* Post-bronchodilator 30%≤FEV1<80% of predicted normal and ost-bronchodilator FEV1/FVC <0.7
* Smoking history of at least 10 pack years

Exclusion Criteria:

* Requiring oxygen therapy on a daily basis
* Exacerbation of airway disease in the 6 weeks prior to screening or between screening and dosing
* Lung reduction surgery
* Respiratory tract infection in the 6 weeks prior to screening
* Significant cardiac history
* History of asthma with onset of symptoms prior to age 40 years
* Active use of certain COPD medications, beta blockers

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Measure: Compare the efficacy of QAX028 at a high dose, as measured by trough forced expiratory volume in 1 second (FEV1), to tiotropium | 7 days treatment

SECONDARY OUTCOMES:
Compare the efficacy of QAX028 at a low dose, as measured by trough FEV1, to tiotropium | 7 days treatment
Measure: Compare the efficacy of QAX028 at two dose levels, as measured by trough FEV1, to placebo | 7 days treatment
Measure: Evaluate the safety and tolerability of two dose levels of QAX028 in COPD patients | 7 days treatment
Measure: Evaluate the pharmacokinetics of multiple inhaled does of QAX028 | 7 days treatment
Measure: Assess bronchodilatory profile, as measured by FEV1, of multiple inhaled doses of QAX028 in COPD patients | 7 days treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Advanced Clinical Research Institute, 1211 W. La Palma Ave, Anaheim, California
  - Sneeze, Wheeze, & Itch Associates, LLC, 2010 Jacobssen Drive, Normal, Illinois
  - Spartanburg Medical Research, 485 Simuel Road, Spartanburg, South Carolina
  - New Orleans Center for Clinical Research - Knoxville, 1928 Alcoa Highway, Knoxville, Tennessee

REFERENCES:
- See also: Results for CQAX028A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5765